CLINICAL TRIAL: NCT06342427
Title: Early Detection of Stomach Cancer With a Liquid Biopsy Based on Exosomal Micro-RNA
Brief Title: Stomach Cancer Exosome-based Detection
Acronym: DESTINEX
Status: Completed | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 23228/DESTINEX
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Gastric Cancer; Gastric Adenocarcinoma; Gastric Cancer Stage; Gastric Neoplasm; Gastric Lesion; Gastric Cancer in Situ; Gastric Cancer Stage IV; Gastric Cancer Stage IIIB; Gastric Cancer Stage III; Gastric Cancer Stage IB; Gastric Cancer Stage IA; Gastric Cancer, Stage 0; Gastric Cancer Stage IIIA; Gastric Cancer Stage II; Gastric Cancer TNM Staging; Gastric Cancer Metastatic to Lung; Gastric Cancer Metastatic to Liver; Gastric Cancer Stage I; Gastric Cancer TNM Staging Primary Tumor (T) T2B
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Formalin-fixed and paraffin-embedded tissue samples Serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients with Gastric Cancer (Training): Individuals with a pathologically confirmed diagnosis of gastric cancer
  Interventions: Diagnostic Test: DESTINEX
- Patients without Gastric Cancer (Training): Individuals without cancer at the time of blood sampling
  Interventions: Diagnostic Test: DESTINEX
- Patients with Gastric Cancer (Validation): Individuals with a pathologically confirmed diagnosis of gastric cancer
  Interventions: Diagnostic Test: DESTINEX
- Patients without Gastric Cancer (Validation): Individuals without cancer at the time of blood sampling
  Interventions: Diagnostic Test: DESTINEX

INTERVENTIONS:
Diagnostic Test: DESTINEX — A panel of microRNA, whose expression level is tested in serum samples.
  Other Names: DESTINEX (DEtection of STomach NEoplasia in circulating eXosomes)

SUMMARY:
Gastric cancer continues to have a poor prognosis primarily due to the inability to detect it in its early stages. This study will develop and validate a blood assay to facilitate the non-invasive detection of gastric cancer.

DETAILED DESCRIPTION:
Gastric cancer continues to have a poor prognosis primarily due to the inability to detect it in its early stages. Because conventional endoscopy is invasive and costly, gastric cancer is currently not considered to be screenable at a population level. However, if one could find less invasive and cheaper tools that accurately detect gastric cancer in its early stages, it could make a significant difference. Accurate biomarkers could help identify patients with gastric cancer before it becomes incurable.

This study aims to develop a non-invasive test to detect gastric cancer early. It consists of four phases:

1. Discovering potential biomarkers with a comprehensive and genome-wide transcriptomic sequencing analysis that will involve gastric cancer tissue, normal tissue, and serum samples from patients with gastric cancer, as well as samples from people without the disease.
2. Using machine learning to develop a combination "signature" of cell-free (cf) and exosomal (exo)-miRNA in serum specimens from a training cohort.
3. A validation of this signature in an independent cohort to confirm its accuracy.
4. An evaluation of the temporal trend of this signature in paired samples collected pre-surgery and post-surgery to investigate their potential and specificity as indicators of minimal residual disease.

In summary, this study aims to develop a highly accurate and cost-effective blood test for detecting gastric cancer early. Success could lead to significant improvements in clinical practice by catching cancer when it is most treatable. By combining different genetic markers (cell-free microRNA and exosomal microRNA) for accuracy, this study has the potential to reduce gastric cancer deaths and could lead to new screening methods in the future.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of stage I, II, III, IV gastric cancer (TNM classification, 8th edition) (cases).
* Received standard diagnostic and staging procedures as per local guidelines, and at least one sample was drawn before receiving any curative-intent treatment.
* Confirmed cancer-free status at the time of study inclusion (Non-disease controls).

Exclusion Criteria:

* Lack of written informed consent.
* Systemic therapy before sampling.
* Synchronous gastric and non-gastric cancer diagnosed at or before surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two cohorts of individuals with and without gastric cancer (cases and controls, respectively)
Sampling Method: Non-Probability Sample
Enrollment: 809 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Sensitivity | Through study completion, an average of 1 year
  True positive rate: the probability of a positive test result, conditioned on the individual truly being positive

SECONDARY OUTCOMES:
Specificity | Through study completion, an average of 1 year
  True negative rate: the probability of a negative test result, conditioned on the individual truly being negative
Proportion of correct predictions (true positives and true negatives) among the total cases (i.e., accuracy) | Through study completion, an average of 1 year
  A measure of trueness: proportion of correct predictions (both true positives and true negatives) among the total number of cases examined

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Goel, PhD, Principal Investigator — City of Hope Medical Center
Locations (3):
- City of Hope Medical Center, Duarte, California, United States
- Japan (2):
  - Nagoya University, Nagoya
  - Mie University, Tsu

IPD SHARING:
Plan to Share IPD: Undecided
Data collected for the study will be made available to others, including de-identified participant data, at publication, via a signed data access agreement and at the discretion of the investigators' approval of the proposed use of such data

REFERENCES:
- [Background] Smyth EC, Nilsson M, Grabsch HI, van Grieken NC, Lordick F. Gastric cancer. Lancet. 2020 Aug 29;396(10251):635-648. doi: 10.1016/S0140-6736(20)31288-5. PMID 32861308
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Nishiwada S, Cui Y, Sho M, Jun E, Akahori T, Nakamura K, Sonohara F, Yamada S, Fujii T, Han IW, Tsai S, Kodera Y, Park JO, Von Hoff D, Kim SC, Li W, Goel A. Transcriptomic Profiling Identifies an Exosomal microRNA Signature for Predicting Recurrence Following Surgery in Patients With Pancreatic Ductal Adenocarcinoma. Ann Surg. 2022 Dec 1;276(6):e876-e885. doi: 10.1097/SLA.0000000000004993. Epub 2021 Jun 16. PMID 34132691
- [Background] Pasechnikov V, Chukov S, Fedorov E, Kikuste I, Leja M. Gastric cancer: prevention, screening and early diagnosis. World J Gastroenterol. 2014 Oct 14;20(38):13842-62. doi: 10.3748/wjg.v20.i38.13842. PMID 25320521
- [Background] Lee JH, Kim JG, Jung HK, Kim JH, Jeong WK, Jeon TJ, Kim JM, Kim YI, Ryu KW, Kong SH, Kim HI, Jung HY, Kim YS, Zang DY, Cho JY, Park JO, Lim DH, Jung ES, Ahn HS, Kim HJ. Clinical practice guidelines for gastric cancer in Korea: an evidence-based approach. J Gastric Cancer. 2014 Jun;14(2):87-104. doi: 10.5230/jgc.2014.14.2.87. Epub 2014 Jun 30. PMID 25061536
- [Background] Shimada H, Noie T, Ohashi M, Oba K, Takahashi Y. Clinical significance of serum tumor markers for gastric cancer: a systematic review of literature by the Task Force of the Japanese Gastric Cancer Association. Gastric Cancer. 2014 Jan;17(1):26-33. doi: 10.1007/s10120-013-0259-5. Epub 2013 Apr 10. PMID 23572188
- [Background] Heitzer E, Haque IS, Roberts CES, Speicher MR. Current and future perspectives of liquid biopsies in genomics-driven oncology. Nat Rev Genet. 2019 Feb;20(2):71-88. doi: 10.1038/s41576-018-0071-5. PMID 30410101
- [Background] Siravegna G, Mussolin B, Venesio T, Marsoni S, Seoane J, Dive C, Papadopoulos N, Kopetz S, Corcoran RB, Siu LL, Bardelli A. How liquid biopsies can change clinical practice in oncology. Ann Oncol. 2019 Oct 1;30(10):1580-1590. doi: 10.1093/annonc/mdz227. PMID 31373349
- [Background] Jung G, Hernandez-Illan E, Moreira L, Balaguer F, Goel A. Epigenetics of colorectal cancer: biomarker and therapeutic potential. Nat Rev Gastroenterol Hepatol. 2020 Feb;17(2):111-130. doi: 10.1038/s41575-019-0230-y. Epub 2020 Jan 3. PMID 31900466
- [Background] Rupaimoole R, Slack FJ. MicroRNA therapeutics: towards a new era for the management of cancer and other diseases. Nat Rev Drug Discov. 2017 Mar;16(3):203-222. doi: 10.1038/nrd.2016.246. Epub 2017 Feb 17. PMID 28209991
- [Background] Schwarzenbach H, Nishida N, Calin GA, Pantel K. Clinical relevance of circulating cell-free microRNAs in cancer. Nat Rev Clin Oncol. 2014 Mar;11(3):145-56. doi: 10.1038/nrclinonc.2014.5. Epub 2014 Feb 4. PMID 24492836
- [Background] Shigeyasu K, Toden S, Zumwalt TJ, Okugawa Y, Goel A. Emerging Role of MicroRNAs as Liquid Biopsy Biomarkers in Gastrointestinal Cancers. Clin Cancer Res. 2017 May 15;23(10):2391-2399. doi: 10.1158/1078-0432.CCR-16-1676. Epub 2017 Jan 31. PMID 28143873
- [Background] Toiyama Y, Okugawa Y, Goel A. DNA methylation and microRNA biomarkers for noninvasive detection of gastric and colorectal cancer. Biochem Biophys Res Commun. 2014 Dec 5;455(1-2):43-57. doi: 10.1016/j.bbrc.2014.08.001. Epub 2014 Aug 13. PMID 25128828
- [Background] Okugawa Y, Grady WM, Goel A. Epigenetic Alterations in Colorectal Cancer: Emerging Biomarkers. Gastroenterology. 2015 Oct;149(5):1204-1225.e12. doi: 10.1053/j.gastro.2015.07.011. Epub 2015 Jul 26. PMID 26216839
- [Background] Nik Mohamed Kamal NNSB, Shahidan WNS. Non-Exosomal and Exosomal Circulatory MicroRNAs: Which Are More Valid as Biomarkers? Front Pharmacol. 2020 Jan 20;10:1500. doi: 10.3389/fphar.2019.01500. eCollection 2019. PMID 32038230
- [Background] Lopez K, Lai SWT, Lopez Gonzalez EJ, Davila RG, Shuck SC. Extracellular vesicles: A dive into their role in the tumor microenvironment and cancer progression. Front Cell Dev Biol. 2023 Mar 21;11:1154576. doi: 10.3389/fcell.2023.1154576. eCollection 2023. PMID 37025182
- [Background] Zhu L, Li J, Gong Y, Wu Q, Tan S, Sun D, Xu X, Zuo Y, Zhao Y, Wei YQ, Wei XW, Peng Y. Exosomal tRNA-derived small RNA as a promising biomarker for cancer diagnosis. Mol Cancer. 2019 Apr 2;18(1):74. doi: 10.1186/s12943-019-1000-8. PMID 30940133
- [Background] Miyazaki K, Wada Y, Okuno K, Murano T, Morine Y, Ikemoto T, Saito Y, Ikematsu H, Kinugasa Y, Shimada M, Goel A. An exosome-based liquid biopsy signature for pre-operative identification of lymph node metastasis in patients with pathological high-risk T1 colorectal cancer. Mol Cancer. 2023 Jan 6;22(1):2. doi: 10.1186/s12943-022-01685-8. PMID 36609320
- [Background] Lane JS, Hoff DV, Cridebring D, Goel A. Extracellular Vesicles in Diagnosis and Treatment of Pancreatic Cancer: Current State and Future Perspectives. Cancers (Basel). 2020 Jun 10;12(6):1530. doi: 10.3390/cancers12061530. PMID 32532129
- [Background] Lennon KM, Wakefield DL, Maddox AL, Brehove MS, Willner AN, Garcia-Mansfield K, Meechoovet B, Reiman R, Hutchins E, Miller MM, Goel A, Pirrotte P, Van Keuren-Jensen K, Jovanovic-Talisman T. Single molecule characterization of individual extracellular vesicles from pancreatic cancer. J Extracell Vesicles. 2019 Nov 4;8(1):1685634. doi: 10.1080/20013078.2019.1685634. eCollection 2019. PMID 31741725
- [Background] Akers JC, Gonda D, Kim R, Carter BS, Chen CC. Biogenesis of extracellular vesicles (EV): exosomes, microvesicles, retrovirus-like vesicles, and apoptotic bodies. J Neurooncol. 2013 May;113(1):1-11. doi: 10.1007/s11060-013-1084-8. Epub 2013 Mar 2. PMID 23456661
- [Background] Chaput N, Thery C. Exosomes: immune properties and potential clinical implementations. Semin Immunopathol. 2011 Sep;33(5):419-40. doi: 10.1007/s00281-010-0233-9. Epub 2010 Dec 21. PMID 21174094
- [Background] Nakamura K, Zhu Z, Roy S, Jun E, Han H, Munoz RM, Nishiwada S, Sharma G, Cridebring D, Zenhausern F, Kim S, Roe DJ, Darabi S, Han IW, Evans DB, Yamada S, Demeure MJ, Becerra C, Celinski SA, Borazanci E, Tsai S, Kodera Y, Park JO, Bolton JS, Wang X, Kim SC, Von Hoff D, Goel A. An Exosome-based Transcriptomic Signature for Noninvasive, Early Detection of Patients With Pancreatic Ductal Adenocarcinoma: A Multicenter Cohort Study. Gastroenterology. 2022 Nov;163(5):1252-1266.e2. doi: 10.1053/j.gastro.2022.06.090. Epub 2022 Jul 16. PMID 35850192
- [Background] Li A, Yu J, Kim H, Wolfgang CL, Canto MI, Hruban RH, Goggins M. MicroRNA array analysis finds elevated serum miR-1290 accurately distinguishes patients with low-stage pancreatic cancer from healthy and disease controls. Clin Cancer Res. 2013 Jul 1;19(13):3600-10. doi: 10.1158/1078-0432.CCR-12-3092. Epub 2013 May 22. PMID 23697990